CLINICAL TRIAL: NCT02457481
Title: An Alternative Culture Medium to Better Support Preimplantation Embryo Development in Vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Foundation for Fertility Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFFR-OEC-2015
Record Dates: First submitted 2015-05-13; First posted 2015-05-29 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Infertility; Reproductive Techniques, Assisted
Keywords: Embryo Culture Techniques; Embryonic Development
MeSH Terms: conditions — Infertility; Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Embryo Culture medium (Experimental): Embryos from each patient are randomly allocated to culture in the commercial or experimental embryo culture medium (half of the embryos in commercial and half in experimental medium).
  Interventions: Device: Embryo Culture medium

INTERVENTIONS:
Device: Embryo Culture medium — Two step sequential embryo culture medium system

SUMMARY:
The purpose of this research study is to evaluate a newly developed embryo culture media system for human clinical use in ART.

DETAILED DESCRIPTION:
Egg retrieval will be performed as per standard operating procedures. Eggs from a single patient are mixed together in a single group during the normal recovery and washing procedure following egg retrieval. The single group of eggs will be divided in half, then the embryologist will randomly place each half into one of the two culture media treatments, commercial or experimental. All mature eggs collected at retrieval will undergo fertilization per standard operating procedures according to physician recommendations. After fertilization (day 0), standard procedures involve in vitro embryo culture in a sequential two step media system. After confirmation of fertilization success on day 1, embryos are cultured until day 3 in step 1 medium (both commercial and experimental media are two step sequential culture systems). On day 3, embryos are evaluated and moved from step one to step two culture medium. On day 5 and day 6, embryo development will be assessed. Good quality blastocysts will either be transferred fresh or cryopreserved for later transfer and/or genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult women of any age who come to Colorado Center for Reproductive Medicine for fertility treatment using IVF.
* Patients can be of any race, culture, sexual orientation or ethnicity.

Exclusion Criteria:

* Minors are excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
embryo development | 7 days after egg retrieval
  Blastocyst development and quality on days 5 and 6 of culture
pregnancy rate | 2 months after egg retrieval
  The incidence of implantation and pregnancy following embryo transfer, including initial pregnancy test and ultrasound examination.
offspring weight | 1 year after egg retrieval
  The birth weight of children born
offspring gender | 1 year after egg retrieval
  The gender of children born

SECONDARY OUTCOMES:
fertilization | 2 days after egg retrieval
  the percentage of mature eggs that successfully fertilized normally
euploid embryos | 1 month after egg retrieval
  For patients undergoing comprehensive chromosome screening, percent normal euploid blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Krisher, PhD, Principal Investigator — NFFR
Locations (2):
- United States (2):
  - Fertility Laboratories of Colorado, Lone Tree, Colorado
  - National Fooundation for Fertility Research, Lone Tree, Colorado